CLINICAL TRIAL: NCT04805450
Title: A Prospective, Randomized, Multicenter Study Comparing Sems Placement With and Without Biliary Sphincterectomy in Patients With Malignant Biliary Obstruction
Brief Title: Sems Placement With and Without Biliary Sphincterectomy in Patients With Malignant Biliary Obstruction
Acronym: SEMS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ES vs noES-1
Record Dates: First submitted 2015-08-18; First posted 2021-03-18 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Malignant Bile Duct Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ES before SEMS placement (Active Comparator): ERCP with ES before biliary fully covered SEMS placement.
  Interventions: Procedure: ES before fully covered SEMS placement
- no ES before SEMS placement (Active Comparator): ERCP without ES before biliary fully covered SEMS placement.
  Interventions: Procedure: no ES before fully covered SEMS placement

INTERVENTIONS:
Procedure: ES before fully covered SEMS placement
  Arms: ES before SEMS placement
Procedure: no ES before fully covered SEMS placement
  Arms: no ES before SEMS placement

SUMMARY:
Placement of biliary self expanding metal stent (SEMS) is indicated when malignant common bile duct obstruction is encountered [1]. Currently, there is still controversy regarding the use of endoscopic sphincterotomy (EST) before the placement of biliary stents [2-5].

The aim of this prospective randomized, multicenter study is to investigate the role of EST before fully covered SEMS placement in patients with neoplastic biliary obstruction.

ELIGIBILITY:
* Inclusion criteria

  * Patients referred for endoscopic retrograde cholangiopancreatography
  * Malignant bile duct obstruction
  * Signed written informed consent
  * Age > 18
* Exclusion criteria

  * Inability to provide inform consent
  * Pregnancy or lactation
  * Suspected perforation of the GI tract
  * Anatomical alterations due to previous surgery (Billroth surgery)
  * Coagulation alterations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1075 (Estimated)
Dates: Start 2015-10-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the need for ES before SEMS placement in patients with malignant bile duct obstruction. | During procedure

SECONDARY OUTCOMES:
To evaluate immediate and delayed post ERCP complications including pancreatitis, SEMS migration, bleeding and perforation. | periprocedural and 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy

REFERENCES:
- [Background] Dumonceau JM, Tringali A, Blero D, Deviere J, Laugiers R, Heresbach D, Costamagna G; European Society of Gastrointestinal Endoscopy. Biliary stenting: indications, choice of stents and results: European Society of Gastrointestinal Endoscopy (ESGE) clinical guideline. Endoscopy. 2012 Mar;44(3):277-98. doi: 10.1055/s-0031-1291633. Epub 2012 Feb 1. PMID 22297801
- [Background] Simmons DT, Petersen BT, Gostout CJ, Levy MJ, Topazian MD, Baron TH. Risk of pancreatitis following endoscopically placed large-bore plastic biliary stents with and without biliary sphincterotomy for management of postoperative bile leaks. Surg Endosc. 2008 Jun;22(6):1459-63. doi: 10.1007/s00464-007-9643-8. Epub 2007 Nov 20. PMID 18027045
- [Background] Artifon EL, Sakai P, Ishioka S, Marques SB, Lino AS, Cunha JE, Jukemura J, Cecconello I, Carrilho FJ, Opitz E, Kumar A. Endoscopic sphincterotomy before deployment of covered metal stent is associated with greater complication rate: a prospective randomized control trial. J Clin Gastroenterol. 2008 Aug;42(7):815-9. doi: 10.1097/MCG.0b013e31803dcd8a. PMID 18285718
- [Background] Giorgio PD, Luca LD. Comparison of treatment outcomes between biliary plastic stent placements with and without endoscopic sphincterotomy for inoperable malignant common bile duct obstruction. World J Gastroenterol. 2004 Apr 15;10(8):1212-4. doi: 10.3748/wjg.v10.i8.1212. PMID 15069728
- [Background] Cui PJ, Yao J, Zhao YJ, Han HZ, Yang J. Biliary stenting with or without sphincterotomy for malignant biliary obstruction: a meta-analysis. World J Gastroenterol. 2014 Oct 14;20(38):14033-9. doi: 10.3748/wjg.v20.i38.14033. PMID 25320543